CLINICAL TRIAL: NCT05019872
Title: Al Dente or Well Done? The Eating Rate of a Pasta Meal Modified by Texture
Acronym: ESPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SEC WUR 2021
Record Dates: First submitted 2021-07-19; First posted 2021-08-25 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Eating Behavior
Keywords: Eating rate; Pasta; Oral Processing; Eating Behaviour; Texture; Hardness
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: All participants receive twelve pasta samples differing in the hardness of carrots and penne, and the addition of sauce
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Penne hard (Active Comparator): 20 g penne cooked for 7 minutes
  Interventions: Behavioral: (Components of) pasta meal
- Penne soft (Active Comparator): 20 g penne cooked for 20 minutes
  Interventions: Behavioral: (Components of) pasta meal
- Carrot hard (Active Comparator): 50 g diced carrot cooked for 2 minutes
  Interventions: Behavioral: (Components of) pasta meal
- Carrot soft (Active Comparator): 50 g diced carrot cooked for 20 minutes
  Interventions: Behavioral: (Components of) pasta meal
- Penne hard + sauce (Active Comparator): 20 g penne cooked for 7 minutes + 10 g tomato sauce
  Interventions: Behavioral: (Components of) pasta meal
- Penne soft + sauce (Active Comparator): 20 g penne cooked for 20 minutes + 10 g tomato sauce
  Interventions: Behavioral: (Components of) pasta meal
- Carrot hard + sauce (Active Comparator): 50 g diced carrot cooked for 2 minutes + 10 g tomato sauce
  Interventions: Behavioral: (Components of) pasta meal
- Carrot soft + sauce (Active Comparator): 50 g diced carrot cooked for 20 minutes + 10 g tomato sauce
  Interventions: Behavioral: (Components of) pasta meal
- Penne hard + carrot hard + sauce (Active Comparator): 20 g penne cooked for 7 minutes + 50 g diced carrot cooked for 2 minutes + 20 g tomato sauce
  Interventions: Behavioral: (Components of) pasta meal
- Penne hard + carrot soft + sauce (Active Comparator): 20 g penne cooked for 7 minutes + 50 g diced carrot cooked for 20 minutes + 20 g tomato sauce
  Interventions: Behavioral: (Components of) pasta meal
- Penne soft + carrot hard + sauce (Active Comparator): 20 g penne cooked for 20 minutes + 50 g diced carrot cooked for 2 minutes + 20 g tomato sauce
  Interventions: Behavioral: (Components of) pasta meal
- Penne soft + carrot soft + sauce (Active Comparator): 20 g penne cooked for 20 minutes + 50 g diced carrot cooked for 20 minutes + 20 g tomato sauce
  Interventions: Behavioral: (Components of) pasta meal

INTERVENTIONS:
Behavioral: (Components of) pasta meal — Samples will be provided one by one in cups labeled with an unique code.

SUMMARY:
Rationale: The world-wide rising obesity rates are a major health problem. Therefore, people should moderate food intake. A lower eating rate will decrease the energy intake. The eating rate of foods can be modified by changing the texture without affecting their acceptability. Harder, chunkier, more viscous, and more voluminous foods will decrease the eating rate and thus energy intake. However, the impact of texture on oral processing has mostly been studied as a model or single food system, whereas a diet consists of many different food products often consumed in combination. Little has been researched on the effect of food texture on eating rate within the context of realistic meals. It is not known if the eating rate of a meal is determined by the eating rate component with the lowest eating rate or if there is an additive effect of the eating rates of all components of the meal.

Objective: The aim of the ESPA study is to determine how the eating rate of a pasta meal can be changed by manipulating the hardness of the ingredients and to investigate if the eating rate of a meal is determined by the eating rate of the component with the lowest eating rate or if there is an additive effect of the eating rates of all components of the meal.

Study design: The study is a randomized crossover trial. All participants receive all pasta samples.

Study population: Healthy adults (n=50) between 18-55 years old with European nationality, and a BMI between 18.5-30 kg/m2.

Intervention: Participants will attend three test sessions during lunch in which in total twelve pasta samples will be consumed. The pasta samples will consists of individual or combined pasta noodles, vegetables, and sauce differing in hardness. The order of the samples will be randomized. After the consumption of the test samples, the participants will rate their appetite and the sensory characteristics of the samples. During the test sessions, participants will be video recorded to determine their eating behavior.

Main study parameters/endpoints: The main study outcome is the eating rate (g/min). Secondary outcomes are the oral processing characteristics assessed with the video recordings (meal duration [min], bite duration [min], number of bites, number of chews, average bite size [g], average amount of chews per bite, and oral sensory exposure time [min]) and sensory characteristics rated on a visual analogue scale (liking [flavor, texture, and overall], flavor intensity, sweetness, saltiness, sourness, hardness, and chewiness).

DETAILED DESCRIPTION:
The study has a randomized crossover design with three test sessions. All participants receive twelve pasta samples (four per test session) and are their own control (within subject effects).

Participants attend three test sessions during which they eat four pasta samples. The pasta samples will have a fixed amount and differ in pasta noodle and vegetable hardness. Eight pasta samples will consist out of only penne or carrots with or without sauce. Four pasta samples will consist out of penne, carrots, and sauce. The sample order will be randomized, but in each test session only one or two of sample 9 to 12 will be served. The samples will be served on a plate together with a fork.

Procedure of the study:

Throughout study period :

* No use of drugs
* Medication use + illness should be reported

Evening preceding test day:

• Not allowed to eat or drink after 22.00 except for water

Morning of test day:

* Do not perform intensive exercise
* Eat the same breakfast at the same time each test day
* If wanted, eat the same morning snack at the same time each test day
* Not allowed to eat or drink two hours prior the study session except for water
* Have a negative corona test

Lunch

* Give instructions (eat as you normally would do, eat the whole sample without taking breaks or sips of water in between, you can take a new bite before you swallowed the previous one)
* Seated at sensory booth with fork, knife, spoon, 200 mL of water and three pieces of a plain cracker
* Question about food consumption that morning
* Appetite questionnaire
* Eat the pasta sample (one of twelve conditions) while recording eating behavior
* Sensory questionnaire
* Appetite questionnaire
* Taste neutralization by waiting for two minutes, taking sip of water and bite of cracker
* Repeat * ... * until four pasta samples are consumed
* Appetite questionnaire

Participants will be recruited from Wageningen and surroundings using an e-mailing list, social media, and flyers. Healthy (self-report), normal weight (18.5-30 kg/m2) men and women between 18-55 years old will be included. Participants need to have European nationality, and have to be able to understand and speak English (self-report), because of the sensory questionnaire and appetite questionnaire which will be in English and have difficult direct translations to Dutch. As 90% of the people that show interest in the study are university students this should not be a problem. The BMI range is based on the average BMI in the Netherlands, which is 25 kg/m2 but around 50% of the Dutch population is overweight. To be able to include sufficient subjects it was therefore chosen to widen the BMI range and include people up to a BMI of 30 kg/m2. Due to the within subject design this will not influence the outcome of the study, but results will be more generalizable to people with an average weight.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-55 years old at the day of inclusion
* European nationality
* Able to understand and speak English fluently or without difficulty (self-report)
* BMI 18.5-30 kg/m2 (self-report)
* Good general health and appetite (self-report)
* Regular consumers of pasta with tomato sauce (commonly once or more per month)

Exclusion Criteria:

* Pregnant or lactating women
* Smoking
* Braces (not including a dental wire) or oral piercing
* Difficulties with swallowing, chewing and/or eating in general
* Suffering from an endocrine or eating disorder, gastrointestinal illness or illness of the thyroid gland, respiratory disease, or diabetes
* Having taste or smell disorders (self-report)
* Use of medication that may influence study outcomes (self-report)
* Consuming on average more than 21 glasses of alcohol per week
* Not willing to stop using drugs during the study period (from inclusion till last test session)
* Intensive exercising more than eight hours per week
* Allergies or intolerance to any ingredient of the test meals
* Don't like pasta with tomato sauce or its ingredients (<five on a nine point Likert scale)
* Men having facial hair such as a beard as facial movements cannot be analyzed
* Signed up for participating in another research study
* Employee of Human Nutrition department of Wageningen university
* Employee, thesis student or intern at the chair group of Sensory Science and Eating Behaviour Human Nutrition or Food Quality and Design (WUR)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Eating rate (g/min) | 1 sample, up to 30 minutes
  Amount of the sample divided by the consumption time of the sample, measured with video recording.

SECONDARY OUTCOMES:
Meal duration (min) | 1 sample, up to 30 minutes
  Time to consume one sample, measured with video recording.
Bite duration (min) | 1 sample, up to 30 minutes
  Measured with video recording.
Number of bites | 1 sample, up to 30 minutes
  Measured with video recording.
Number of chews | 1 sample, up to 30 minutes
  Measured with video recording.
Average bite size (g) | 1 sample, up to 30 minutes
  Measured with video recording.
Chews per bite | 1 sample, up to 30 minutes
  Measured with video recording.
Oro-sensory exposure time (min) | 1 sample, up to 30 minutes
  Measured with video recording.
Liking flavour | 1 sample, up to 30 minutes
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Liking texture | 1 sample, up to 30 minutes
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Liking overall | 1 sample, up to 30 minutes
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Sweetness | 1 sample, up to 30 minutes
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Saltiness | 1 sample, up to 30 minutes
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Sourness | 1 sample, up to 30 minutes
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Hardness | 1 sample, up to 30 minutes
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Chewiness | 1 sample, up to 30 minutes
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line

CONTACTS AND LOCATIONS:
Overall Officials: Lise AJ Heuven, MSc, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Human Nutrition Department, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No